CLINICAL TRIAL: NCT01239069
Title: A Phase II, Prospective, Randomized, Observer-masked, Parallel-group, Multi-center Study Assessing the Safety and Efficacy of Two Concentrations Compared to Placebo for the Treatment of Dry Eye Disease
Brief Title: Safety and Efficacy Study of DE-110 Ophthalmic Suspension for the Treatment of Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30-002
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- DE-110 ophthalmic suspension high dose (Experimental)
  Interventions: Drug: DE-110 ophthalmic suspension high dose
- DE-110 ophthalmic suspension low dose (Experimental)
  Interventions: Drug: DE-110 ophthalmic suspension low dose
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DE-110 ophthalmic suspension high dose — ophthalmic suspension; high dose; QID
  Arms: DE-110 ophthalmic suspension high dose
Drug: DE-110 ophthalmic suspension low dose — ophthalmic suspension; low dose; QID
  Arms: DE-110 ophthalmic suspension low dose
Other: Placebo — DE-110 ophthalmic suspension vehicle;QID
  Arms: Placebo

SUMMARY:
Investigate the Safety and Efficacy of Two Concentrations of DE-110 Compared to Placebo for the Treatment of Dry Eye Disease

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of dry eye
* Not wear contact lenses during study
* 18 years or older
* Understand and provide written consent
* Negative pregnancy test and use acceptable method of contraception

Exclusion Criteria:

* Use of any topical ocular medication
* Any type of ocular surgery
* Diagnosis of on-going ocular infection and/or allergic conjunctivitis
* Uncontrolled systemic conditions/lid abnormalities
* Corneal transplants
* Females who are pregnant, nursing or planning a pregnancy
* Participation in another drug trial concurrently or within 30 days prior to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of DE-110 | 12 weeks

SECONDARY OUTCOMES:
Individual Response Rate | 12 weeks
Individual Efficacy | 12 weeks
Individual Symptoms | 12 weeks

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Inglewood, California
  - Newport Beach, California
  - Petaluma, California
  - Torrance, California
  - Bloomfield, Connecticut
  - Bradenton, Florida
  - Brooksville, Florida
  - Largo, Florida
  - Rosewell, Georgia
  - Louisville, Kentucky
  - Bangor, Maine
  - Cleveland, Ohio
  - San Antonio, Texas
  - Norfolk, Virginia